CLINICAL TRIAL: NCT03605654
Title: A Phase 2/3, Prospective, Randomized, Multi-center, Open-Label, Controlled Trial to Assess the Efficacy & Safety of Cellular Immunotherapy With MDR-102 for Induction of Immune Quiescence™in Recipients of HLA-mismatched, LD Kidney Transplants
Brief Title: Cellular Immunotherapy in Recipients of Human Leukocyte Antigen (HLA)-Mismatched, Living Donor Kidney Transplants
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Medeor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDR-102-mMLK
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Immunosuppressive Agents; Adrenal Cortex Hormones; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Intervention Model Description: A low-dose Total Lymphoid Irradiation and anti- thymocyte globulin combined with a single infusion of MDR-102
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Arm (Experimental): A low-dose Total Lymphoid Irradiation and anti- thymocyte globulin combined with a single infusion of MDR-102 post-kidney transplant and standard anti-rejection medications in recipients of 1, 2, or 3 out of 6 human leukocyte antigen (HLA)-mismatched, living donor kidney transplants
  Interventions: Biological: MDR-102
- Active Control Arm (Active Comparator): Standard anti-rejection medications that would be given to kidney transplant recipients who are outside the study
  Interventions: Drug: Immunosuppressive Agents
- Non-Randomized Exploratory Arm (Experimental): A low-dose Total Lymphoid Irradiation and anti- thymocyte globulin combined with a single infusion of MDR-102 post-kidney transplant and standard anti-rejection medications in recipients of 4, 5, or 6 out of 6 human leukocyte antigen (HLA)-mismatched, living donor kidney transplants
  Interventions: Biological: MDR-102

INTERVENTIONS:
Biological: MDR-102 — Enriched CD34+ hematopoietic stem cells and defined dose of CD3+ T-cells
  Arms: Investigational Arm; Non-Randomized Exploratory Arm
Drug: Immunosuppressive Agents — Standard Anti-Rejection Medications that would be given to kidney transplant recipients who are outside the study
  Other Names: Corticosteroids; Mycophenolate Mofetil; Tacrolimus
  Arms: Active Control Arm

SUMMARY:
The Phase 2 primary objective is to evaluate achievement of persistent mixed chimerism and withdrawal of at least one immunosuppression drug for a minimum of 6 months with no episodes of biopsy-proven acute rejection or transplant kidney loss induced by cellular immunotherapy with MDR-102 in recipients of 1, 2, or 3 out of 6 human leukocyte antigen (HLA)-mismatched, living donor kidney transplants.

The Phase 3 primary objective is to evaluate achievement of induction of immune quiescence by cellular immunotherapy with MDR-102 in recipients of 1, 2, or 3 out of 6 HLA-mismatched, living donor kidney transplants. Immune quiescence is defined as remaining on maintenance immunosuppression monotherapy with Tac or CsA for 12 months or more after completion of anti-rejection immunosuppression drug therapy reduction with no episodes of biopsy-proven acute rejection, transplant kidney loss, or subject deat.

DETAILED DESCRIPTION:
Currently, patients receiving a transplanted kidney are required to take life-long immunosuppressive medications to prevent rejection of the transplanted kidney. These medications carry substantial side effects. In addition, these medicines often do not completely control damage to the kidney from the recipients' immune system, ultimately causing the kidney to fail.

Medeor Therapeutics is developing a novel cell-based therapy as personalized cellular immunotherapies to improve outcomes in organ transplant recipients.

The purpose of the current Phase 2/3 study is to demonstrate the efficacy and safety of MDR-102 for the induction of immune quiescence in a prospective, randomized, open-label, multi-center clinical trial. MDR-102 is intended to induce mixed lymphohematopoietic chimerism and donor specific immune quiescence in order to preserve transplant kidney function, avert transplant kidney rejection, and reduce the cumulative and serious side effects associated with immunosuppression drugs.

ELIGIBILITY:
Inclusion Criteria:

* Recipient Inclusion Criteria:

  * Planned recipient of a first kidney allograft from an human leukocyte antigen (HLA)-matched, living related donor. Zero-mismatch transplants are excluded
  * Age ≥18 and ≤65 years
  * Single solid organ recipient (kidney only)
  * ABO compatibility with donor
* Donor Inclusion Criteria:

  * Human leukocyte antigen (HLA)-mismatched first degree (parent, child or sibling) or second-degree (child of a sibling) relative of the prospective recipient participant. Zero-mismatch transplants are excluded
  * Age ≥18 and ≤65 years
  * Prepared to be a living related kidney donor, and capable of undergoing granulocyte-colony stimulating factor (G-CSF) mobilization and apheresis of hematopoietic cells

Exclusion Criteria:

* Recipient Exclusion Criteria:

  * Underlying kidney disease with a high risk of disease recurrence in the transplanted kidney
  * Baseline positive donor-specific anti-HLA antibody testing
  * Is taking immunosuppressive therapy
  * Prior hematopoietic cell transplant, organ transplant, any cell therapy, or any gene therapy
  * Evidence of prior hepatitis B (HBV) or hepatitis C (HCV)
* Donor Exclusion Criteria:

  * History of autoimmune disorders
  * History of type 1 or type 2 diabetes mellitus
  * Tests confirmed positive for human immunodeficiency virus (HIV), HBV, HCV
  * History of infection with Zika virus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phase 2 Primary Outcome: Achievement of persistent mixed chimerism and withdrawal of at least one Immunosuppression drug for a minimum of 6 months | 6 months
  Persistent mixed chimerism is defined as:
  • At least 6 months of persistent white blood cells mixed chimerism consisting of at least 5% donor white blood cells in whole blood or in at least one white blood cells lineage
Phase 3 Primary Outcome: proportion of subjects achieving immune quiescence | 24 months
  Immune quiescence is defined as:
  * Achievement of the required duration of persistent donor mixed chimerism (i.e., 6 months) to permit mycophenolic acid drug (e.g., mycophenolate mofetil) immunosuppression stoppage without a taper at approximately 12 months post-kidney transplant surgery,
  * Successful stoppage of mycophenolic acid drug (e.g., mycophenolate mofetil) at 12 + 1 months post-kidney transplant surgery, and
  * Subsequent successful maintenance on calcineurin inhibitor monotherapy for at least 12 additional months (out to at least 24 months post-kidney transplant surgery) without biopsy-proven acute rejection, transplant kidney loss, or subject death

CONTACTS AND LOCATIONS:
Overall Officials: Lenuta Micsa, MD, Study Director — Medeor Therapeutics

IPD SHARING:
Plan to Share IPD: Undecided